CLINICAL TRIAL: NCT02139137
Title: Evaluating a Novel Working Memory Training Program to Decrease Symptoms of PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rick Gulizia (Other)
Responsible Party: Sponsor-Investigator, Rick Gulizia, Director of Research Affairs, San Diego State University
Organization: San Diego State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F31MH088170 (NIH)
Record Dates: First submitted 2014-05-12; First posted 2014-05-15 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Interference Control Condition (Experimental): Computerized training program requiring participants to repeatedly practice controlling interference on a cognitive task
  Interventions: Other: Computerized Cognitive Training - active
- Low Interference Control Condition (Active Comparator): Computerized training program requiring participants to minimally practice controlling interference on a cognitive task
  Interventions: Other: Computerized cognitive training - sham

INTERVENTIONS:
Other: Computerized Cognitive Training - active — Cognitive training using working memory span task
  Arms: High Interference Control Condition
Other: Computerized cognitive training - sham — Sham training condition
  Arms: Low Interference Control Condition

SUMMARY:
The study is designed to evaluate the effect of a novel computer training program on PTSD.

DETAILED DESCRIPTION:
Post-traumatic stress Disorder (PTSD) is a chronic and debilitating disorder that affects millions of people each year (Kessler et al., 2005). Although effective psychosocial and pharmacological treatments exist for this disorder, as many as 50 percent of individuals still experience symptoms after treatment (Schottenbaeur et al., 2008). Empirical literature suggests that cognitive deficits may play a role in maintaining symptoms in individuals with PTSD through a variety of mechanisms, including decreased cognitive control over intrusive thoughts (Verwoerd et al., in press) and dysregulation in neural circuitry linking prefrontal cognitive control functions and amygdala activity (McNally, 2007). The goals of the proposed research are to improve the candidate's understanding of cognitive mechanisms of PTSD symptoms while building skills in conducting treatment research. The application aims to test a novel methodology for approaching PTSD treatment based on modification of underlying cognitive mechanisms of the disorder. To this end, 50 participants with PTSD will be randomly assigned to an 8-session executive control training condition designed to improve working memory functioning or a control condition. The aims of this study are 1) To test the effect of a working memory training program on working memory performance and 2) To examine the effects of this program on PTSD symptoms. The research plan is complemented by a set of training goals for the candidate to achieve over the proposed award period. These include 1) training in the use of fMRI and neuropsychological assessment 2) additional coursework and seminars in cognitive science and biostatistics for use in future work, 3) experience with teaching in the undergraduate and graduate setting and presenting original work for publication in preparation for a career in academic research. Taken together, the research and training components of this grant application will facilitate the candidate's long-term goal of conducting treatment outcome and basic mechanism research in PTSD. Moreover, as per the strategic plan outlined by NIMH, this application is designed develop an innovative intervention based on prior clinical research and knowledge of cognitive and neurobiological features of the disorder, and will advance knowledge of mechanisms of fear learning. It is designed to target core cognitive features of the disorder in an effort to reduce symptoms. PUBLIC HEALTH RELEVANCE: Post-traumatic stress disorder impacts millions of Americans, and is associated with significant personal distress as well as societal cost. The current application is designed to examine the effect of a novel working memory training program on PTSD symptoms. This approach is promising in that it may be a cost- effective and accessible method for decreasing symptoms associate with this disorder.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-65
* Primary DSM-IV diagnosis of PTSD secondary to sexual trauma

Exclusion Criteria:

* Current trauma or PTSD-focused psychosocial treatment
* Active suicidality, evidence of substance dependence in the past 6 months
* Evidence of current or past schizophrenia
* Bipolar disorder
* Organic mental disorder

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-01; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Bomyea, M.S., Principal Investigator — San Diego State University/University of California, San Diego; Ariel J Lang, Ph.D., Principal Investigator — University of California, San Diego

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bomyea J, Stein MB, Lang AJ. Interference control training for PTSD: A randomized controlled trial of a novel computer-based intervention. J Anxiety Disord. 2015 Aug;34:33-42. doi: 10.1016/j.janxdis.2015.05.010. Epub 2015 Jun 10. PMID 26114901

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 47 individuals consented to participate in the study. Of those, 42 started the study and were randomized. The remaining 5 were not assigned to either condition. Intent to treat analyses are presented using last observation carried forward for all continuous measures.
Period: Overall Study
Arm/Group | High Interference Control Condition | Low Interference Control Condition
Started | 22 | 20
Completed | 15 | 10
Not Completed | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Interference Control Condition | Low Interference Control Condition | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 20 | 42
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician Administered PTSD Scale; Re-experiencing
Description: Model estimations of the means and standard deviation of posttreatment score at the mean level of baseline severity reported below.
  Scale range: 0-40, higher values indicate greater symptom severity
Time Frame: Baseline, Week 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | High Interference Control Condition | Low Interference Control Condition
Number analyzed (Participants) | 22 | 20
units on a scale | 11.78 (1.14) | 15.69 (1.20)

2. Secondary Outcome: Clinician Administered PTSD Scale Total Score - Responder Status
Description: Number of Participants Who Responded According to Clinician Administered PTSD Scale Total Score
Time Frame: Week 4
Population: Number of participants analyzed is based on the number of participants who completed the post-treatment CAPS interview.
Measure: Count of Participants; unit: Participants
Arm/Group | High Interference Control Condition | Low Interference Control Condition
Number analyzed (Participants) | 13 | 8
Participants | 11 | 6

3. Secondary Outcome: Change in Depression: Beck Depression Inventory
Description: Scale Range: 0-63; higher scores indicate greater symptom severity
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Interference Control Condition | Low Interference Control Condition
Number analyzed (Participants) | 22 | 20
units on a scale | 6.8 (8.9) | 4.6 (8.9)

4. Secondary Outcome: Change in General Anxiety: Spielberger State-Trait Anxiety Inventory
Description: Range: 20-80; higher scores indicate greater symptom severity
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Interference Control Condition | Low Interference Control Condition
Number analyzed (Participants) | 22 | 20
units on a scale | 6.1 (8.6) | 3.0 (9.3)

5. Secondary Outcome: Change in Functional Impairment; Sheehan Disability Scale
Description: Range: 0-30; greater values indicate greater disability severity ratings
Time Frame: Baseline, Week 4
Population: Data at one time point for one participant in the LIC condition are not available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Interference Control Condition | Low Interference Control Condition
Number analyzed (Participants) | 22 | 19
units on a scale | 3.2 (7.2) | 1.7 (6.3)

ADVERSE EVENTS:
Arm/Group | High Interference Control Condition | Low Interference Control Condition
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No